CLINICAL TRIAL: NCT02885597
Title: Juanbi Pill Combined With Methotrexate for Rheumatoid Arthritis: Multi-center Random Controlled Clinical Trials
Brief Title: Juanbi Pill for Rheumatoid Arthritis
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cui xuejun (Other)
Collaborators: Shanghai Yueyang Integrated Medicine Hospital (Other); Longhua Hospital (Other); Shanghai Guanghua Hospital of Integrated Traditional Chinese and Western Medicine (Other)
Responsible Party: Sponsor-Investigator, Cui xuejun, Director, Shanghai University of Traditional Chinese Medicine
Organization: Shanghai University of Traditional Chinese Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Juanbi pill
Record Dates: First submitted 2016-08-18; First posted 2016-08-31 (Estimated); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: Juanbi Pill; Rheumatoid Arthritis
Keywords: Juanbi Pill; Methotrexate; Active; Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid; Motor Activity | interventions — Methotrexate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Juanbi group (Experimental): participants should administrate both Juanbi pill and Methotrexate
  Interventions: Drug: Juanbi pill; Drug: Methotrexate
- placebo group (Placebo Comparator): participants should administrate both Juanbi pill placebo and Methotrexate
  Interventions: Drug: Juanbi pill placebo; Drug: Methotrexate

INTERVENTIONS:
Drug: Juanbi pill — 4g, twice a day, 3month, oral
  Other Names: Experimental: Juanbi group
  Arms: Juanbi group
Drug: Juanbi pill placebo — 4g, twice a day, 3month, oral
  Other Names: Placebo Comparator: placebo group
  Arms: placebo group
Drug: Methotrexate — 5mg, once a week, 3 month, oral
  Other Names: Experimental: Juanbi group; Placebo Comparator: placebo group

SUMMARY:
The purpose of this study is to determine whether Juanbi Pill combined with methotrexate are effective in the treatment of active Rheumatoid Arthritis (RA).

DETAILED DESCRIPTION:
Rheumatoid arthritis patients are suffering from painful and swelling of joints as well as joint destruction and functional disability with the duration of disease activity. Patients and physician try to find a way to alleviate the swell and tenderness of joints to avoid irreversible joints impairment, for evidence indicating that early aggressive treatment results in greater improvement than therapy initiated later in the disease course.

As a complementary and alternative medicine (CAM), herbal medicines have the potential to achieve a clinical remission, or push the disease back to low disease activity. In traditional Chinese medicine (TCM), rheumatoid arthritis is a Bi syndrome and Juanbi decotion (notopterygium root, radix angelicae pubescentis, Gentiana macrophylla, Kadsura Pepper Stem, Mulberry Twig, Angelica sinensis, Ligusticum wallichii, frankincense, Radix Aucklandiae, shaved cinnamon barka and liquorice ) is a medicine specially for Bi syndrome and it has been used in Chinese for hundreds of years. Juanbi pill is the raw extration of Juanbi decotion for the sake of convenience of quality control and storage.

Although the long term usage of Juanbi decotion, there is no high quality evidence about the decotion on rheumatoid arthritis. Using a well-designed clinical trial, the investigators will survey the effectiveness of concurrent use of this decotion in relieving disease activity. Therefore, the present study is to examine effectiveness and safety of Juanbi Pill, a compound traditional Chinese herbal medicine on rheumatoid arthritis in a randomized, double-blind, placebo-controlled trial. Results of this study will provide evidence regarding the value of the Juanbi pill as an intervention to lower the disease activity and protect the affected joints from deformity.

ELIGIBILITY:
Inclusion Criteria:

* Adults with rheumatoid arthritis (score more then 5 of ACR (American College Of Rheumatology) /EULAR (European League Against Rheumatism), 2009 )
* moderate-to-severe disease activity (Disease Activity Score for 28-joint counts (DAS28) of more than 3.2
* an onset of symptoms within 12 months before enrollment, no prior exposure to more than 10mg oral glucocorticoids or biologic agents
* paid employment or unpaid but measurable work (e.g., caring for a family and home)

Exclusion Criteria:

* combined with other disease such as adjuvant arthritis, lupus arthritis, osteoarthritis and et al.
* abnormal liver and my kidney function
* pregnancy or have a plan of pregnancy,breast feeding women
* severe chronic or acute disease interfering with therapy attendance
* alcohol or substance abuse

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-07 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Rate of ACR (American College Of Rheumatology) 50 | at 3 months
changes of The Disease Activity Score (DAS) 28 | from baseline to 3 months
changes of the van der Heijde modified Sharp score | from baseline to 12 months

SECONDARY OUTCOMES:
changes of The Disease Activity Score (DAS) 28 | from baseline to 2 weeks
changes of The Disease Activity Score (DAS) 28 | from baseline to 1 month
changes of The Disease Activity Score (DAS) 28 | from baseline to 6 months
changes of The Disease Activity Score (DAS) 28 | from baseline to 12 months
Rate of ACR(American College Of Rheumatology)50 | at 2 weeks
Rate of ACR(American College Of Rheumatology)50 | at 1 month
Rate of ACR(American College Of Rheumatology)50 | at 2 months
Rate of ACR(American College Of Rheumatology)50 | at 6 months
Rate of ACR(American College Of Rheumatology)50 | at 12 months
change score of Health Assessment Questionnaire - Disability Index | from baseline to 2 weeks
change score of Health Assessment Questionnaire - Disability Index | from baseline to 1 month
change score of Health Assessment Questionnaire - Disability Index | from baseline to 2 months
change score of Health Assessment Questionnaire - Disability Index | from baseline to 3 months
change score of Health Assessment Questionnaire - Disability Index | from baseline to 6 months
change score of Health Assessment Questionnaire - Disability Index | from baseline to 12 months
change score of Patient Assessment of Arthritis Pain | from baseline to 2 weeks
change score of Patient Assessment of Arthritis Pain | from baseline to 1 month
change score of Patient Assessment of Arthritis Pain | from baseline to 2 months
change score of Patient Assessment of Arthritis Pain | from baseline to 3 months
change score of Patient Assessment of Arthritis Pain | from baseline to 6 months
change score of Patient Assessment of Arthritis Pain | from baseline to 12 months
change score of Patient Global Assessment of Arthritis | from baseline to 2 weeks
change score of Patient Global Assessment of Arthritis | from baseline to 1 month
change score of Patient Global Assessment of Arthritis | from baseline to 2 months
change score of Patient Global Assessment of Arthritis | from baseline to 3 months
change score of Patient Global Assessment of Arthritis | from baseline to 6 months
change score of Patient Global Assessment of Arthritis | from baseline to 12 months
change score of 36-item Short-Form Health Survey Questionnaire | form baseline to 2 weeks
change score of 36-item Short-Form Health Survey Questionnaire | form baseline to 1 month
change score of 36-item Short-Form Health Survey Questionnaire | form baseline to 2 months
change score of 36-item Short-Form Health Survey Questionnaire | form baseline to 3 months
change score of 36-item Short-Form Health Survey Questionnaire | form baseline to 6 months
change score of 36-item Short-Form Health Survey Questionnaire | form baseline to 12 months
change score of AIS Sleep Scale | from baseline to 2 weeks
change score of AIS Sleep Scale | from baseline to 1 month
change score of AIS Sleep Scale | from baseline to 2 months
change score of AIS Sleep Scale | from baseline to 3 months
change score of AIS Sleep Scale | from baseline to 6 months
change score of AIS Sleep Scale | from baseline to 12 months
rate of ACR20 | at 2 weeks
rate of ACR20 | at 1 month
rate of ACR20 | at 2 months
rate of ACR20 | at 3 months
rate of ACR20 | at 6 months
rate of ACR20 | 12 months
rate of ACR70 | at 2 weeks
rate of ACR70 | at 1 month
rate of ACR70 | at 2 months
rate of ACR70 | at 3 months
rate of ACR70 | at 6 months
rate of ACR70 | at 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Longhua Hospital, Shanghai University of TCM, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Jia QY, Wang YR, Sun DW, Mao JC, Xue L, Gu XH, Yu X, Piao XM, Xu H, Liang QQ. Efficacy and Safety of Juan Bi Pill with Add-on Methotrexate in Active Rheumatoid Arthritis: A 48-Week, Multicentre, Randomized, Double-Blind, Placebo-Controlled Trial. Chin J Integr Med. 2025 Feb;31(2):99-107. doi: 10.1007/s11655-024-3768-7. Epub 2024 Dec 21. PMID 39707138
- [Derived] Wang Q, Wang YR, Jia QY, Liu L, Xu CQ, Wang XY, Yao M, Cui XJ, Shi Q, Wang YJ, Liang QQ. The efficacy of the traditional Chinese medicine Juanbi pill combined with methotrexate in active rheumatoid arthritis: study protocol for a randomized controlled trial. Trials. 2018 Mar 20;19(1):188. doi: 10.1186/s13063-018-2555-1. PMID 29558967